CLINICAL TRIAL: NCT05176015
Title: Randomized Controlled Trial on Nystagmus Assessment for Patients Consulting for Acute Vertigo in the Emergency Department With/Without Frenzel Lens With/Without Form: A Pilot Study
Brief Title: Nystagmus Assessment for Patients Consulting in the Emergency Department for Acute Vertigo
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Pierre La Rochelle, Chief Investigator, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MP-CIBSSSBSL-2021-03
Record Dates: First submitted 2021-10-19; First posted 2022-01-04 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Nystagmus, Acquired; Stroke, Acute
Keywords: nystagmus; stroke; neuroimaging; cardiovascular disease; benign positional paroxystic vertigo
MeSH Terms: conditions — Nystagmus, Pathologic; Stroke; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Frenzel Lens with Diagnostic Algorithm (Experimental): Frenzel lens will be applied on patients' eyes during different diagnostic maneuvers to assess if a nystagmus is present and if present describe its main characteristic.
  Without mentioning to patient, the emergency physician will use a diagnostic algorithm inspired from the TiTrATE approach to interpret the nystagmus and propose the need or the irrelevance for neuro-imaging
  Interventions: Device: Frenzel Lens; Diagnostic Test: Diagnostic Algorithm
- Frenzel Lens without Diagnostic Algorithm (Experimental): Frenzel lens will be applied on patients' eyes during different diagnostic maneuvers to assess if a nystagmus is present and describe its main characteristics. No diagnostic algorithm will be used to interpret nystagmus.
  Interventions: Device: Frenzel Lens
- No Frenzel Lens with Diagnostic Algorithm (Experimental): Nystagmus assessment in different manoeuvres is performed without the use of Frenzel lens.
  Without mentioning to patient, the emergency physician will use a diagnostic algorithm inspired from the TiTrATE approach to interpret the nystagmus and propose the need or the irrelevance for neuro-imaging
  Interventions: Diagnostic Test: Diagnostic Algorithm
- No Frenzel Lens and No Diagnostic Algorithm (No Intervention): The emergency physician is performing the assessment of nystagmus and its interpretation as usual. The Frenzel lens and the diagnostic algorithm are not used.

INTERVENTIONS:
Device: Frenzel Lens — pair of magnifying glasses (+20 dioptres) that are worn by the patient and an illuminating system. On using Frenzel goggles, the nystagmus is better seen as a result of eyes being magnified and inhibition of visual fixation.
  Arms: Frenzel Lens with Diagnostic Algorithm; Frenzel Lens without Diagnostic Algorithm
Diagnostic Test: Diagnostic Algorithm — A diagnostic algorithm using the TiTrate approach: continuous, Intermittent, trigger or spontaneous.
  The diagnostic algorithm use the REDCap software that include different videos to illustrate diagnostic tests and nystagmus types. Different maneuvers: HINTS+ battery, Dix-Hallpike test, Supine Roll test.
  Different Particle Repositioning Techniques will be proposed according to specific tests: Epley and Gufoni maneuvers.
  Risk Score is used to assess stroke risk for transient ischaemic attack (TIA): ABCD2 and the Canadian TIA Risk Score
  Arms: Frenzel Lens with Diagnostic Algorithm; No Frenzel Lens with Diagnostic Algorithm

SUMMARY:
This pilot study is perfomed to validate and document faisability of the use of Frenzel lens and the use of a diagnostic algorithm for the assessment of a special sign (nystagmus) observe in the eyes of patients consulting in the emergency department (ED) for an acute episode of vertigo/dizziness/imbalance.

DETAILED DESCRIPTION:
This pilot study is a randomized controlled trial 2 by 2 design to allocated randomly the Frenzel lens and the diagnostic algorithm. There is no use of sham lens. The usual care opposed to the diagnostic algorithm will be questioned only on the perception of nystagmus by the clinician and the use of repositioning particles technique. The only blinding will be the patients about the use of the algorithm and the outcomes assessor about the use or not of Frenzel lens and the use or not of the diagnostic algorithm.

ELIGIBILITY:
Inclusion Criteria:

* New episode of acute vertigo/dizziness/imbalance occuring during the 28 last days
* Must be able to consent.

Exclusion Criteria:

* No traumatic context before symptoms onset
* No intoxication context
* Glycemia ≤ 3,0 mmol/L
* Only one participation is permitted
* Not able to speak adequately in French or English.
* Reachable for 3 month follow-up

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Nystagmus detection per participant | Day 0
  During eye examination, nystagmus will be characterized according to prominent direction of the fast phase (patients' left, patients' right, up, down, rotational),with their clinical setting or trigger. Overall rate of nystagmus detection by participant. (Rate of typical nystagmus for benign paroxysmal positional vertigo in the Dix-Hallpike maneuver or Supine Head Roll Test. Rate of nystagmus detection in the initial physical exam)

SECONDARY OUTCOMES:
Emergency Department Length of stay | Day 0, from triage time to Emergency Department departure (admission or home discharge)
  Time spent at the emergency department from triage to time of departure for hospital admission or for home discharge assessed up to 48 hours
Rate of neuro-imaging per participant | From day 0 to 12 weeks
  Any imaging to investigate acute intra-cerebral lesion and/or the neck/brain vascular. anomaly : computed tomography imaging; computed tomography angiogram; magnetic resonance angiography; magnetic resonance imaging, vascular neck ultrasound imaging.
Rate of acute stroke per participant | From day 0 to 12 weeks
  Any acute stroke, hemorrhagic or ischemic, diagnosed by neuro-imaging: computed tomography or magnetic resonance imaging
Rate of symptomatic central lesion per participant | From day 0 to 12 weeks
  Any central lesion diagnosed by computed tomography or magnetic resonance imaging that may be related to the initial presentation of vertigo/dizziness/imbalance
Rate of specialised consultations for vertigo/dizziness/imbalance per participant | From day 0 to 12 weeks
  Any specialised consultations (neurology, ear nose and throat (ENT), cardiology or similar) to investigate the acute vertigo/dizziness/imbalance with the final diagnosis. Sumarisation of final diagnosis.
Rate of acute vertigo/dizziness/imbalance related hospitalisation per participant | From day 0 to 12 weeks
  Admission to hospital directly related to vertigo/dizziness/imbalance may be immediate to initial visit or delayed.
Rate of subsequent Emergency Department Visit for Vertigo/dizziness/imbalance per participant | From day 0 t0 12 weeks
  Return visit to the emergency department for vertigo/dizziness/imbalance as chief complaint.
Rate of New Atrial Fibrillation | From day 0 to 12 weeks
  Atrial fibrillation detected by the initial visit electrocardiogram or by long-term cardiac rhythm monitoring (Holter or loop recorder).
Rate of New Stroke at 12 weeks | At 12 weeks
  A stroke free status will be assessed by a validated questionnaire by telephone at tree months and all specialised consultations and neuroimaging will be reviewed for acute stroke diagnosis,
Rate of the use of Particles Repositioning Technique | Day 0
  Once Paroxysmal Positional Vertigo diagnosis is being diagnosed with the Dix-Hallpike test or with the Supine Head Roll test, the use of particles repositioning technique, Epley or Gufoni maneuvers, will be noted with their immediate impact on acute vertigo.
Rate of Emergency Department Visit Return for Benign Paroxysmal Positional Vertigo according to Typical Nystagmus | From day 0 to 12 weeks
  Rate of Emergency Department Visit Return for Benign Paroxysmal Positional Vertigo according to Typical Nystagmus: direction, duration
Initial managment self appreciation of patient presenting in the ED for an acute episode of vertigo/dizziness/imbalance | Day 0
  Simple question answered on a likert scale at the end of the ED encounter. 0% worst, 100% best appreciation.
Adverse Events | From day 0 to 12 weeks
  Combination of stroke, death, neurosurgery, intervenional neuroradiology, thrombolytic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Pierre La Rochelle, MD, MSc, Principal Investigator — Universite Laval
Locations (5):
- Canada (5):
  - Centre Hospitalier d'Amqui, Amqui, Quebec
  - Centre Hospitalier de Matane, Matane, Quebec
  - Centre Hospitalier de Montmagny, Saint Thomas de Montmagny, Quebec
  - Hopital St-Georges, Saint-Georges, Quebec
  - Hopital Notre-Dame-de-Fatima, Ste. Anne de la Pocatière, Quebec

IPD SHARING:
Plan to Share IPD: No